CLINICAL TRIAL: NCT01078363
Title: ACE Inhibition and Cardiac Allograft Vasculopathy
Brief Title: Angiotensin Converting Enzyme (ACE) Inhibition and Cardiac Allograft Vasculopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: VA Palo Alto Health Care System (U.S. Federal Agency); Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, William Fearon, Associate Professor of Medicine, Stanford University
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Prevention
Other Study IDs: SU-12162009-4562; 16155 (William Fuller Fearon)
Record Dates: First submitted 2010-02-26; First posted 2010-03-02 (Estimated); Results first posted 2016-07-27 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2016-12

CONDITIONS: Cardiac Allograft Vasculopathy
Keywords: Heart Transplantation
MeSH Terms: interventions — Ramipril

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ramipril (Active Comparator): ramipril, 5mg starting dose to maximum dose of 20mg daily dose for one year.
  Interventions: Drug: ramipril
- Placebo (Placebo Comparator): Sugar pill manufactured to mimic ramipril 5mg starting dose , increasing to 20mg daily for one year.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ramipril — Use of a ACE ( angiotension converting enzyme) inhibitors post heart Transplant for Blood pressure control.
  Other Names: Altace
  Arms: ramipril
Drug: Placebo — Use of a placebo post heart Transplant for Blood pressure control.
  Arms: Placebo

SUMMARY:
Cardiac transplantation is the ultimate treatment option for patients with end stage heart failure.

Cardiac allograft vasculopathy remains a leading cause of morbidity and mortality after transplantation.

Angiotensin converting enzyme inhibitors are used in less than one half of transplant recipients. Preliminary data suggest that angiotensin converting enzyme inhibitors retard the atherosclerotic plaque development that is the hallmark of cardiac allograft vasculopathy. Moreover, this class of drug appears to increase circulating endothelial progenitor cell number and has anti-inflammatory properties, both of which improve endothelial dysfunction, the key precursor to the development of cardiac allograft vasculopathy.

The objective of this project is to investigate the role of an angiotensin converting enzyme inhibitor, ramipril, in preventing the development of cardiac allograft vasculopathy. During the first month after cardiac transplantation subjects will undergo coronary angiography with intravascular ultrasound measurements of plaque volume in the left anterior descending coronary artery. Using a coronary pressure wire, epicardial artery and microvascular physiology will be assessed. Finally, endothelial function and mediators of endothelial function, including circulating endothelial progenitor cells, will be measured. Subjects will then be randomized in a double blind fashion to either ramipril or placebo. After 1 year, the above assessment will be repeated. The primary endpoint will be the development of cardiac allograft vasculopathy based on intravascular ultrasound-derived parameters. The second aim will be to assess the effect of ramipril on endothelial dysfunction early after transplantation. The final aim is to determine the impact of ramipril on coronary physiology early after transplantation.

DETAILED DESCRIPTION:
During the first 4 years of this study, we plan to recruit patients within the first month after OHT. As has become routine at Stanford, study subjects will undergo baseline coronary angiography and IVUS assessment of their left anterior descending coronary artery. Coronary endothelial function will be assessed as well transmyocardial levels of ADMA and other mediators of endothelial function. Blood samples will be obtained for analyzing circulating EPC number and function. Epicardial and microvascular coronary physiology in the left anterior descending coronary artery will be determined by measuring FFR and IMR with a coronary pressure wire(in the adults only). Subjects will then be randomized to either the ACE I(Ramipril), or to placebo, in addition to their usual medications. During years 2 through 5 of this project, study subjects will undergo the above routine invasive assessments at 1 year after OHT. During the 5th year of this project, data analysis and manuscript preparation will occur.

Table 2. Patient Flowchart Time post OHT Event 0-4 Weeks Recruitment and enrollment 4-6 Weeks Baseline angiogram, endothelial function, coronary physiology and IVUS studies 4-6 (at time of baseline)Weeks Baseline blood sampling for circulating EPC studies 4-6 Weeks Randomization to ramipril or placebo to begin one week after baseline studies 5-7 Weeks Titration up of ramipril or placebo Month 3 and month 6: blood sampling for EPC studies. 11-13 Months 1 year angiogram, endothelial function, coronary physiology and IVUS studies 11-13 Months 1 year blood sampling for circulating EPC studies The primary endpoint of the study will be change in plaque volume as determined by IVUS analysis at baseline and 1 year later, between those treated with ramipril compared to those treated with placebo.

Secondary endpoints will include change in circulating EPC number and function, change in ADMA levels,change in coronary endothelium-dependent vasodilation, and change in coronary physiology (FFR and IMR)from baseline to 1 year. Although there are multiple potential mechanisms by which ACE I might reduce CAV, evaluating each of these is beyond the scope of this project. For this reason, we will focus on the likely common final pathway of endothelial dysfunction mediated by dysregulation of ADMA and NOS, as well as changes in EPCs. If this study shows a benefit to ACE I therapy in this population, the goal of future studies will be to determine the exact mechanism by which this occurs and to perform a large, multicenter study comparing ACE I to placebo with hard clinical endpoints. Study visits include two major time points 1) baseline angiogram and IVUS which include recording of angiographic data, lab data, clinical data. 2)assessment at the usual follow up periods post transplant, and these data points will also be collected for research purposes. after base line which usually occurs one month post transplant plus or minus 2 weeks. F/u = q 2 weeks until two months out from tx, then once per month until six months out from TX, then every two months until the patient is 12 months out from TX. Each routine f/u visit includes a physical exam,vital signs, echocardiogram, chest x-ray, a complete metabolic panel ( contains a Creatinine), Complete blood count, immunosuppressant drug blood levels, and a heart biopsy (at the same intervals described above).

ELIGIBILITY:
Inclusion Criteria:

* Heart transplant recipient within the first month of transplant;
* 12 years of age or older;
* Must have a serum creatinine less than 2.0 mg/dl;
* Will provide written informed consent;
* Female patients of childbearing potential must have negative pregnancy test;
* For pediatric patient, parent(s) will provide consent and the child will sign assent.

Exclusion Criteria:

* Less than 12 years of age;
* Have more than one solid organ transplant at time of heart transplant;
* Has serum creatinine greater than 2.0 mg/dl;
* Pregnancy.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2009-06; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William F Fearon, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - VA Palo Alto Health Care System, Palo Alto, California
  - Stanford University School of Medicine, Stanford, California

REFERENCES:
- [Derived] Arashi H, Sato T, Kobashigawa J, Luikart H, Kobayashi Y, Okada K, Sinha S, Honda Y, Yeung AC, Khush K, Fearon WF. Long-term clinical outcomes with use of an angiotensin-converting enzyme inhibitor early after heart transplantation. Am Heart J. 2020 Apr;222:30-37. doi: 10.1016/j.ahj.2020.01.003. Epub 2020 Jan 9. PMID 32007823
- [Derived] Fearon WF, Okada K, Kobashigawa JA, Kobayashi Y, Luikart H, Sana S, Daun T, Chmura SA, Sinha S, Cohen G, Honda Y, Pham M, Lewis DB, Bernstein D, Yeung AC, Valantine HA, Khush K. Angiotensin-Converting Enzyme Inhibition Early After Heart Transplantation. J Am Coll Cardiol. 2017 Jun 13;69(23):2832-2841. doi: 10.1016/j.jacc.2017.03.598. PMID 28595700
- [Derived] Lee JH, Okada K, Khush K, Kobayashi Y, Sinha S, Luikart H, Valantine H, Yeung AC, Honda Y, Fearon WF. Coronary Endothelial Dysfunction and the Index of Microcirculatory Resistance as a Marker of Subsequent Development of Cardiac Allograft Vasculopathy. Circulation. 2017 Mar 14;135(11):1093-1095. doi: 10.1161/CIRCULATIONAHA.116.025268. No abstract available. PMID 28289008

RESULTS

PARTICIPANT FLOW:
Groups:
- Ramipril: ramipril, 5mg starting dose to maximum dose of 20mg daily dose for one year.
  ramipril or placebo: Use of a ACE ( angiotension converting enzyme) inhibitors versus placebo post heart Transplant for Blood pressure control.
- Placebo: Sugar pill manufactured to mimic ramipril 5mg starting dose , increasing to 20mg daily for one year.
  ramipril or placebo: Use of a ACE ( angiotension converting enzyme) inhibitors versus placebo post heart Transplant for Blood pressure control.
Period: Overall Study
Arm/Group | Ramipril | Placebo
Started | 47 | 49
Completed | 47 | 49
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ramipril | Placebo | Total
Number analyzed (Participants) | 47 | 49 | 96
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (15) | 52 (17) | 53 (16)
Gender [Count of Participants; unit: Participants]
  Female | 11 | 17 | 28
  Male | 36 | 32 | 68

OUTCOME MEASURES:

1. Primary Outcome: Cardiac Allograft Vasculopathy(CAV) Defined as Change in IVUS-assessed Plaque Volume From Baseline to One Year
Description: also called transplant coronary artery disease or cardiac transplant vasculopathy defined as coronary artery stenosis(narrowing) ranging from 30 to 70 percent by coronary angiography. Measured in this study as change in IVUS-assessed Plaque Volume from baseline to one year.
Time Frame: Baseline and 1 Year
Measure: Mean (Standard Deviation); unit: mm3/mm
Arm/Group | Ramipril | Placebo
Number analyzed (Participants) | 47 | 49
mm3/mm | 3.39 (1.65) | 3.65 (1.89)

2. Secondary Outcome: Percentage of Participants With ≥20% Coronary Artery Diameter Reduction After Acetylcholine
Description: The percent change in diameter of the left anterior descending artery was measured by quantitative angiography after acetylcholine and compared to baseline angiography. The percentage of participants who had ≥20% coronary artery diameter reduction after acetylcholine at one year is presented.
Time Frame: At Baseline and 1 Year
Population: Only a subset of participants (those adult patients enrolled at Stanford University) underwent the acetylcholine measurements.
Measure: Number; unit: percentage of participants
Arm/Group | Ramipril | Placebo
Number analyzed (Participants) | 25 | 22
percentage of participants | 9.4 | 4.8

3. Secondary Outcome: ADMA Level at One Year Post Transplant
Description: asymmetric dimethylarginine (ADMA), is an inhibitor of endothelial nitric oxide synthase which is a primary regulator of endothelial function.
Time Frame: 1 year post Transplant
Population: Blood samples were not acquired in all participants which accounts for the discrepancy in number of participants analyzed.
Measure: Mean (Standard Deviation); unit: micromole
Arm/Group | Ramipril | Placebo
Number analyzed (Participants) | 41 | 40
micromole | .54 (.14) | .55 (.16)

4. Secondary Outcome: The Percentage of Endothelial Progenitor Cells ( EPC) in Peripheral Blood in Patients One Year After Transplant
Description: The determination of the percentage of EPC in peripheral blood involved surface staining peripheral blood mononuclear cells (PBMCs) with appropriate fluorescently-labeled antibodies to delineate EPCs from other blood cells, followed by analysis by conventional flow cytometry.
Time Frame: at one year
Population: Not all blood samples obtained were adequate for EPC determination which explains the discrepancy in number of participants analyzed.
Measure: Mean (Standard Deviation); unit: percentage of EPC
Arm/Group | Ramipril | Placebo
Number analyzed (Participants) | 40 | 40
percentage of EPC | .104 (.068) | .098 (.133)

5. Secondary Outcome: Fractional Flow Reserve (FFR) at One Year Post Transplant
Description: FFR is a technique used in coronary catheterization to measure pressure differences across a coronary artery stenosis (narrowing, usually due to atherosclerosis) to determine the likelihood that the stenosis impedes oxygen delivery to the heart muscle (myocardial ischemia). It is defined as the ratio of the distal coronary pressure to the proximal coronary pressure.
Time Frame: at one year post Transplant
Population: Only a subset of participants (adult patients enrolled at Stanford University) underwent fractional flow reserve assessment.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Ramipril | Placebo
Number analyzed (Participants) | 26 | 23
Ratio | .88 (.04) | .90 (.04)

6. Secondary Outcome: Index of Microcirculatory Resistance at One Year Post Heart Transplant
Description: The index of microcirculatory resistance (IMR) is a pressure-temperature sensor guidewire-based measurement, performed during cardiac catheterization, of the minimum microcirculatory resistance in a specific coronary artery. The IMR provides a quantitative measure of coronary microvasculature status.
Time Frame: one year
Population: Only a subset of participants (adult patients enrolled at Stanford University) underwent index of microcirculatory resistance assessment.
Measure: Mean (Standard Deviation); unit: mmHg x seconds
Arm/Group | Ramipril | Placebo
Number analyzed (Participants) | 26 | 22
mmHg x seconds | 14.4 (6.3) | 21.5 (20)

ADVERSE EVENTS:
Arm/Group | Ramipril | Placebo
Serious Adverse Events (participants affected / at risk) | 2/47 | 2/49
Other Adverse Events (participants affected / at risk) | 0/47 | 0/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ramipril (N=47) | Placebo (N=49)
Death (Cardiac disorders) | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No